CLINICAL TRIAL: NCT00046605
Title: Inflammation Genomics and Atherosclerosis - Ancillary to CARDIA
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, David Siscovick, Professor, Medicine, University of Washington
Other Study IDs: 21795; R01HL071017-05 (NIH)
Record Dates: First submitted 2002-09-30; First posted 2002-10-01 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Coronary Arteriosclerosis; Inflammation; Heart Diseases; Thrombosis
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Coronary Artery Disease; Inflammation; Heart Diseases; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To examine the associations of common variation in inflammation/thrombosis genes with intermediate quantitative phenotypes and subclinical coronary atherosclerosis in the Coronary Artery Risk Factor Development in Young Adults (CARDIA) Study, a large, bi-racial cohort study.

DETAILED DESCRIPTION:
BACKGROUND:

Atherosclerosis is a major determinant of coronary heart disease and is determined by the interplay of genetic and environmental risk factors. Although atherosclerosis tends to aggregate in families, it does not exhibit classical Mendelian segregation. Thus, the genes that determine an individual's risk of atherosclerosis likely involve multiple sites within genes and interactions between genes, all of which define a genetic risk that is modified by the host environment.

DESIGN NARRATIVE:

The genetic epidemiology study examines the associations of common variation in inflammation/thrombosis genes with intermediate quantitative phenotypes and subclinical coronary atherosclerosis in the Coronary Artery Risk Factor Development in Young Adults (CARDIA) Study, a large, bi-racial cohort study. The set of 25 candidate genes involve pathways (cytokines, chemokines, and their receptors; cellular adhesion molecules; and, coagulation proteins) and include several receptor-ligand pairs. Using cladistic analysis and the resources of the Program in Genomic Applications (PGA), the investigators will identify a limited set of single nucleotide polymorphisms (range 3-10 SNPs per gene) that characterize common haplotypes in these candidate genes within persons of African descent and European descent. DNA from the CARDIA Year 10 examination (n = 3,950 subjects) will be genotyped for the selected variants that characterize the common haplotypes. Data on the presence of common variants and haplotypes will be incorporated into the CARDIA Study database. Levels of two important intermediate phenotypes, fibrinogen and C-reactive protein (CRP) were previously determined. Non-invasive assessment of coronary atherosclerosis, defined as the presence of coronary artery calcification (CAC), was obtained on CARDIA participants at the Year 15 exam. Analyses will be stratified by race/ethnicity and focus on the associations of the common haplotypes with fibrinogen, CRP, and CAC measured in early adult life. Secondarily, the investigators will explore possible gene-gene and gene-environment interactions. The proposed multi-disciplinary collaboration should enhance the sensitivity and specificity of efforts to assess the associations of common variation in sets of inflammation/thrombosis candidate genes and cardiovascular risk in young adults.

ELIGIBILITY:
Cardiac cohort participants with DNA

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Same as eligibility criteria
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2002-08; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Siscovick, Principal Investigator — University of Washington

REFERENCES:
- [Background] Carlson CS, Aldred SF, Lee PK, Tracy RP, Schwartz SM, Rieder M, Liu K, Williams OD, Iribarren C, Lewis EC, Fornage M, Boerwinkle E, Gross M, Jaquish C, Nickerson DA, Myers RM, Siscovick DS, Reiner AP. Polymorphisms within the C-reactive protein (CRP) promoter region are associated with plasma CRP levels. Am J Hum Genet. 2005 Jul;77(1):64-77. doi: 10.1086/431366. Epub 2005 May 16. PMID 15897982